CLINICAL TRIAL: NCT07066982
Title: A Phase 1/2 Open-Label, Multicenter Trial of Sequential Infusion of CD146-Targeted and HER2-Targeted CAR T Cells in Patients With Advanced Sarcomas
Brief Title: Sequential Infusion of CD146-Targeted and HER2-Targeted CAR T Cells in Patients With Advanced Sarcomas
Acronym: BAH2573-103
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essen Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBI202571-103
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma; Sarcoma, Kaposi; Sarcoma, Ewing; Sarcoma,Soft Tissue; Sarcoma of Bone and Connective Tissue; Sarcoma, Synovial; Sarcoma Metastatic; Sarcomas, Germinoblastic; Sarcoma of Bone
Keywords: Sarcoma; CD146; HER2; CAR-T; Sarcoma of Bone
MeSH Terms: conditions — Sarcoma; Sarcoma, Kaposi; Sarcoma, Ewing; Osteosarcoma; Sarcoma, Synovial; Lymphoma

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this clinical trial will receive a carefully designed treatment regimen. Before the infusion of HER2 and CD146 CAR-T cells, participants will undergo preconditioning chemotherapy. This chemotherapy serves to create an optimal environment for CAR-T cell therapy to effectively target and eliminate Cancer cells. Following chemotherapy, participants will receive the infusion of CD146 and HER-2 CAR-T cells.
Masking Description: Open-label clinical trials are a category of clinical research where the masking is minimal or nonexistent. In such trials, both the participants and the researchers are fully aware of the treatment assignments, which means participants know the treatment they are receiving, and researchers are aware of each participant's treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD146/HER2 CAR T cells, chemotherapy (Experimental): Patients will be administered fludarabine phosphate intravenously (IV) over a 30-minute period on days -4 to -2. Additionally, cyclophosphamide will be administered intravenously (IV) over 60 minutes on day -2. Subsequently, patients will receive CD146 HER-2 CAR T cells intravenously (IV) over a duration of 10-20 minutes on day 0. Patients who exhibit positive responses to the initial dose of CD146/HER2 CAR T cells, do not experience unacceptable side effects, and have a sufficient quantity of cells available may be eligible to receive 2 or 3 additional doses of CD146/HER2 CAR T cells.
  Interventions: Biological: CD146/HER2 CAR-T cells

INTERVENTIONS:
Biological: CD146/HER2 CAR-T cells — The intervention in this clinical trial involves a novel approach using CD146/HER2 Chimeric Antigen Receptor T (CAR T) cells combined with chemotherapy. The goal is to assess safety and efficacy in patients with specific hematologic malignancies.
  Treatment Regimen:
  Patients in the trial will undergo the following regimen:
  Fludarabine Phosphate (Days -4 to -2): IV administration of fludarabine phosphate over 30 minutes on days -4 to -2. It's part of the preparatory regimen to enhance the body's response to CAR T-cell therapy.
  Cyclophosphamide (Day -2): IV cyclophosphamide over 60 minutes on day -2.
  BCMA/GPRC5D Chimeric Antigen Receptor T Cells (Day 0): IV administration of investigational therapy, CD146/HER-2 CAR T cells, over 10-20 minutes on day 0.
  Additional Doses: Eligible patients responding well to the initial CD146/HER-2 CAR-T cell infusion without unacceptable side effects and sufficient CAR-T cell availability may receive 2 or 3 additional doses.

SUMMARY:
This is an open-label, non-randomized, multicenter Phase 1/2 trial evaluating a dual CAR-T cell therapy targeting CD146 and HER2 in patients with advanced sarcoma. Participants will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine, followed by sequential infusion of autologous CD146-specific and HER2-specific CAR-T cells. The Phase 1 portion will employ a dose-escalation design to assess safety and determine the recommended Phase 2 dose, while the Phase 2 expansion will evaluate preliminary efficacy (tumor response and survival outcomes). Approximately 40 patients (children and adults) with relapsed or refractory sarcomas will be enrolled across multiple centers. All participants will be followed for up to 36 months to monitor dose-limiting toxicities, objective response rates, progression-free survival, overall survival, and long-term safety.

DETAILED DESCRIPTION:
Advanced sarcomas have poor prognoses with existing treatments, and novel immunotherapies are needed. HER2 is expressed in subsets of sarcomas (e.g. osteosarcoma), and a Phase 1 trial of HER2-targeted CAR T cells in sarcoma demonstrated that this approach is tolerable and can induce objective responses. However, in that study the median progression-free survival was only ~2.4 months and 1-year progression-free survival rate was ~21%, highlighting the need for enhanced efficacy. CD146 (MCAM) is a cell adhesion molecule highly expressed in many solid tumors (including sarcomas) and on tumor vasculature. Overexpression of CD146 is implicated in tumor progression and metastasis, so immunotherapy against CD146 is a promising strategy to inhibit metastatic spread. Dual targeting of HER2 and CD146 may therefore broaden anti-tumor activity by addressing tumor heterogeneity and the tumor microenvironment, potentially improving response durability.

Study Design: This trial consists of two phases. The Phase 1 portion is a dose-escalation (3+3 design) of sequential CD146 CAR-T and HER2 CAR-T cell infusions to evaluate safety, identify dose-limiting toxicities (DLTs), and determine the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) for each CAR-T product when given sequentially. In Phase 1, small cohorts of patients will receive escalating doses of the CAR-T cells; safety data will be reviewed by a monitoring committee before dose progression. Once the RP2D is established, the trial will expand into Phase 2. The Phase 2 portion is a dose-expansion at the RP2D, treating a larger cohort of patients to evaluate preliminary efficacy and further characterize safety at that dose.

All enrolled participants will undergo lymphodepletion with cyclophosphamide (e.g. 500-1000 mg/m²/day for 2 days) and fludarabine (e.g. 30 mg/m²/day for 3-5 days) prior to CAR-T cell infusion, per standard CAR-T therapy protocols. Following lymphodepletion, patients will receive sequential infusions of two investigational CAR-T cell products: first an infusion of CD146-targeted CAR T cells, then an infusion of HER2-targeted CAR T cells. (The interval between the two CAR-T infusions may be on the same day or consecutive days, as defined in the protocol, to allow for safe administration of both products in sequence.) This sequential dual-CAR-T approach is intended to attack the tumor on two fronts: targeting CD146-expressing elements of the tumor and vasculature, as well as HER2-expressing tumor cells.

Endpoints and Follow-Up: Patients will be closely monitored for acute toxicities, including cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS), which are known risks with CAR-T therapies. The primary endpoints focus on safety: incidence of DLTs within the first cycle (e.g. 28 days post-CAR T infusion) and the establishment of an MTD/RP2D. Secondary endpoints include measures of anti-tumor efficacy: objective response rate (ORR) per RECIST 1.1 or appropriate sarcoma response criteria, progression-free survival (PFS), overall survival (OS), and duration of response. Immune correlates (such as CAR T cell expansion and persistence, cytokine levels, and tumor biopsy analyses) will be explored to understand the mechanism of response or resistance.

Participants will be followed for up to 36 months after CAR-T administration. This long-term follow-up allows assessment of durable responses, late relapses, and delayed adverse events. Safety follow-up will include periodic physical exams, laboratory tests, and imaging. Responses will be assessed at regular intervals (e.g. every 8-12 weeks) using imaging (MRI/CT) to evaluate tumor size. Long-term monitoring will also watch for potential delayed toxicities such as late-onset cytopenias or secondary malignancies. The trial's multi-center design will facilitate the enrollment of a diverse patient population and ensure robust collection of safety and efficacy data. The ultimate goal is to determine whether the sequential infusion of CD146 and HER2 directed CAR T-cells can be safely administered and show sufficient anti-sarcoma activity to warrant further clinical development. Essen Biotech, as the sponsor, will oversee regulatory compliance, data collection, and analysis in alignment with GCP and ClinicalTrials.gov reporting requirements.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival time ≥3 months;
* Diagnosis: Histologically or cytologically confirmed sarcoma (soft tissue or bone sarcoma), that is metastatic, locally advanced, or refractory to standard therapy. This may include osteosarcoma, Ewing sarcoma, rhabdomyosarcoma, leiomyosarcoma, or other high-grade sarcomas. Patients must have evidence of measurable disease as per RECIST or applicable criteria.
* Prior Treatment: Patients should have received and progressed on or not be candidates for standard first-line treatments. There is no limit on number of prior lines of therapy, but at least one prior systemic therapy for sarcoma is typically required (unless no standard therapy exists for the subtype). A minimum wash-out period (e.g. 2 weeks) from previous treatments (chemotherapy, radiation, or other immunotherapy) is required before lymphodepletion.
* Age and Performance Status: Participants age 12 years and older (both adolescent and adult patients are eligible; for minors, legal guardian consent is required). Upper age limit of ~75 years, or as determined by medical fitness. ECOG performance status 0-1 (or Karnofsky ≥70% for pediatric patients), indicating subjects are ambulatory and able to perform light work.
* Organ Function: Adequate organ function to undergo cytotoxic chemotherapy and cell transfer therapy, including: cardiac ejection fraction ≥50%; baseline oxygen saturation >92% on room air; adequate bone marrow reserves (absolute neutrophil count ≥1.0×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥8 g/dL), hepatic function (e.g. bilirubin ≤1.5× ULN, AST/ALT ≤2.5× ULN), and renal function (e.g. creatinine clearance ≥50 mL/min or age-appropriate normal).
* Tumor Antigen Expression: Expression of CD146 and/or HER2 in the tumor is recommended (as assessed by immunohistochemistry or flow cytometry on a tumor sample). Note: At least one of the target antigens (CD146 or HER2) should be present on the tumor; if feasible, patients should have tumor tissue tested for these markers. (In cases where testing is unavailable, enrollment may proceed based on histology known to often express these targets, per investigator judgment.)
* Consent: Ability to understand and provide written informed consent (or assent for minors with consent of legal guardian). Patients (or guardians) must be willing to comply with trial procedures and follow-up.

Exclusion Criteria:

* Recent Therapies: Prior treatment with any CAR-T cell therapy or other gene-modified T-cell therapy is excluded. Also exclude patients who received any investigational drug, immunotherapy (e.g. checkpoint inhibitor), or major surgery within a certain interval (e.g. 4 weeks) prior to enrollment. Concurrent enrollment in another interventional clinical trial is not allowed.
* Recent Therapies: Prior treatment with any CAR-T cell therapy or other gene-modified T-cell Infections: Active uncontrolled infection, including active hepatitis B or C infection, or HIV infection with uncontrolled viral load. Patients must not have evidence of active tuberculosis or other severe infections. All patients will be screened for HBV, HCV, and HIV at baseline.
* Immunosuppression: Use of systemic immunosuppressive medications (such as chronic corticosteroids at >10 mg prednisone daily or equivalent) within 7 days prior to leukapheresis. (Physiologic replacement doses of steroids are permitted.) Patients with a history of allogeneic stem cell transplant or solid organ transplant are excluded (due to the need for immunosuppression and risk of graft-versus-host or graft rejection).
* Medical Comorbidities: Any significant uncontrolled medical condition that would, in the investigator's judgment, make the patient an unsuitable candidate for CAR-T therapy. For example: active autoimmune diseases requiring immunosuppression, clinically significant heart failure (NYHA class III-IV), unstable angina or myocardial infarction within 6 months, severe chronic respiratory disease requiring supplemental oxygen, or psychiatric conditions that would interfere with study participation and follow-up.
* Pregnancy/Breastfeeding: Women who are pregnant or breastfeeding are excluded due to unknown risks of the treatment to a fetus or infant. Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use effective contraception during the study and for a suitable period after CAR-T infusion (e.g. 1 year), given the potential for sustained CAR T-cell activity. A negative serum pregnancy test is required for females of childbearing potential before starting lymphodepletion.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD19/BCMA chimeric antigen receptor (CAR) T cells | 28 days
  Will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 at three dose levels until the maximum tolerated dose (MTD) is determined.

SECONDARY OUTCOMES:
Rate of successful manufacture and expansion of the CD146/HER-2 chimeric antigen receptor (CAR) T cells | 60 days
  satisfy the targeted dose level and meet the required release specifications outlined in the Certificate of Analysis (COA)

CONTACTS AND LOCATIONS:
Locations (1):
- District One Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No